CLINICAL TRIAL: NCT06390761
Title: Acupuncture for the Treatment of Parkinson's Disease Related Constipation
Brief Title: Efficacy of Acupuncture for the Treatment of Parkinson's Disease Related Constipation
Acronym: AFPDC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFPDC; 2020qn06 (Other Grant/Funding Number: Xi'an Health Commission Research Project)
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease; Constipation; Non-motor Symptom; Randomized Controlled Trial
MeSH Terms: conditions — Parkinson Disease; Constipation | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Acupuncture Group (Experimental): The intervention is going to be executed using the acupoints EX-HN1（Sishencong),LI4 (Hegu),ST25 (Tianshu),ST37(Shangjuxu),ST36(Zusanli),ST44 (Neiting), ST44 (Taichong), SP6 (Sanyinjiao) and CV4 (Shuangyuan).The acupuncture needles will be inserted to a depth of 0.8 to 1 cm in the acupuncture group.
  Interventions: Procedure: Acupuncture
- The Sham Acupuncture Group (Sham Comparator): The sham acupuncture group's needles will be inserted to a depth of 0.2 to 0.3 cm with nonacupuncture points located 0.5 cm in lateral to the real acupoint or to the right for midline points.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — All acupoints were selected based on traditional Chinese medicine theory and previous articles on PD and constipation.

SUMMARY:
The purpose of the study is to evaluate the efficacy of acupuncture in treating Parkinson's disease related constipation (PDC). In the randomized controlled clinical trial study, patients meeting the criteria for inclusion will be randomly enrolled and divided into two groups in a 1:1 ratio: the acupuncture group and the sham acupuncture group. The intervention is going to be executed using the acupoints EX-HN1（Sishencong),LI4 (Hegu),ST25 (Tianshu),ST37(Shangjuxu),ST36(Zusanli),ST44 (Neiting), ST44 (Taichong), SP6 (Sanyinjiao) and CV4 (Shuangyuan).The acupuncture needles will be inserted to a depth of 0.8 to 1 cm in the acupuncture group. The sham acupuncture group's needles will be inserted to a depth of 0.2 to 0.3 cm with nonacupuncture points located 0.5 cm in lateral to the real acupoint or to the right for midline points. During the study, researchers will observe changes in complete spontaneous bowel movements (CSBMs), Constipation Symptom and Efficacy Assessment Scale (CSEAS) (including the six dimensions of difficulty, Bristol, time, incompleteness, frequency,and bloating), the Patient-Assessment of Constipation Quality of Life questionnaire (PAC-QOL), and the Unified Parkinson's Disease Rating Scale (UPDRS) at baseline (week 0), post-treatment (week 4), and follow-up (week 12).Colonic transit time measurement and conventional anorectal manometry were evaluated at the above time points.

DETAILED DESCRIPTION:
Age, sex, duration of disease, and equivalent daily dose of levodopa were assessed at baseline. From the beginning of the baseline phase to the end of the follow-up phase, patients were requested to complete an electronic bowel diary, which was supervised by an independent outcome assessor. The primary outcome in this study was the number of weekly CSBMs. Weekly CSBMs were collected at baseline (week 0), post-treatment (week 4), and follow-up (week 12), and differences from baseline levels were compared at week 4 and week 12. Anorectal manometry (AM) and colonic transit time (TT) were assessed in the two groups using standardized procedures. In brief, for TT evaluation, patients swallowed a capsule containing 24 radiopaque markers. Abdominal radiographs from patients in the erect posture were acquired 5 days after markers intake. During the test period, patients were instructed to maintain their habitual diet and to avoid laxatives, enema and suppositories. According to manufacturer's indications, the TT was described as "normal" if at least 19 markers (80%) were expelled at day 5. The AM was performed using the stationed pull-through technique, with a 4-channel water-perfused catheter linked to an electronic manometer. The catheter was inserted via the anal canal and positioned in the rectum, with the patient in a left-lateral decubitus position. Functional parameters included the resting and squeeze pressures, the ability of the anal sphincter to relax with straining, the recto-anal inhibitory reflex (RAIR) and the rectal sensation.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of PD (according to the Movement Disorder Society's revised clinical diagnostic criteria for Parkinson's disease in 2015) and functional constipation (according to the Rome IV diagnostic criteria) ;
2. Age between 35 and 80 years;
3. Hoehn-Yahr grade ≤ 3;
4. No medications taken within 2 weeks that may affect gastrointestinal function (such as prucalopride and probiotics);
5. No anticipation in other clinical trials within 1 month;
6. Voluntary engagement in this study, ability to sign the informed consent, and cooperation in the completion of the bowel diary and scale filling.

Exclusion Criteria:

1. Organic lesions of the digestive system (such as intestinal adhesions, obstructions, tumors, or malformations in the gastrointestinal tract);
2. A history of abdominal or anorectal surgery that may affect intestinal transit, systemic diseases that may affect the dynamics of the digestive tract (such as diabetes and hyperthyroidism);
3. Serious life-threatening diseases (such as severe cardiovascular diseases and malignant tumors);
4. Skin lesions that were inappropriate for needling, the viscose allergy that prevented acupuncture device attachment;
5. Pregnant or lactating women.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of weekly CSBMs | Weekly CSBMs were collected at baseline (week 0), post-treatment (week 4), and follow-up (week 12), and differences from baseline levels were compared at week 4 and week 12.
  Complete spontaneous bowel movements

SECONDARY OUTCOMES:
Constipation Symptom and Efficacy Assessment Scale (CSEAS) | CSEAS were collected at baseline (week 0), post-treatment (week 4), and follow-up (week 12), and differences from baseline levels were compared at week 4 and week 12.
  Including the six dimensions of difficulty, Bristol, time, incompleteness, frequency, and bloating
Patient-Assessment of Constipation Quality of Life questionnaire (PAC-QOL) | PAC-QOL were collected at baseline (week 0), post-treatment (week 4), and follow-up (week 12), and differences from baseline levels were compared at week 4 and week 12.
  To assess quality of life in patients with constipation. It includes questions about the impact of constipation symptoms on the daily life of the patient, such as difficult defecation, bloating, abdominal pain, etc.
The Unified Parkinson's Disease Rating Scale (UPDRS) | These were assessed at baseline (week 0), post-treatment (week 4), and follow-up (week 12), and differences from baseline levels were compared at week 4 and week 12.
  To assess the severity and symptoms
TT | TT was assessed at baseline (week 0), post-treatment (week 4), and follow-up (week 12), and differences from baseline levels were compared at week 4 and week 12.
  Colonic transit time
AM | AM was assessed at baseline (week 0), post-treatment (week 4), and follow-up (week 12), and differences from baseline levels were compared at week 4 and week 12.
  Anorectal manometry

CONTACTS AND LOCATIONS:
Overall Officials: Gejuan Zhang, Doctor, Study Director — The dean
Locations (1):
- Xi 'an No.3 Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Data is managed by the project team and can be shared according to individual needs